CLINICAL TRIAL: NCT06679374
Title: Reducing Falls With Varenicline in Hypocholinergic Parkinson Disease
Acronym: CRANE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vikas Kotagal (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor-Investigator, Vikas Kotagal, Associate Professor of Neurology, University of Michigan
Organization: University of Michigan (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HUM00254213; 1UG3NS133515-01A1 (NIH)
Record Dates: First submitted 2024-11-05; First posted 2024-11-07 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-03

CONDITIONS: Parkinson Disease
Keywords: Mild Cognitive impairment; Multitasking; Reduce falls; Hypocholinergic
MeSH Terms: conditions — Parkinson Disease; Cognitive Dysfunction | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind study. The study personnel (except for select staff at the Data Coordinating Center (DCC) and research pharmacy).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Varenicline (Experimental)
  Interventions: Drug: Varenicline

INTERVENTIONS:
Drug: Placebo — Participants will take one pill (.5 milligrams) a day for days 1-3 and then one pill (.5 milligrams) in the morning and one pill in the evening days 4-30 and months 2-12. In month 13 participants will take one pill in the morning days 1-3. Participants will be off study drug month 13 days 4-30.
  Arms: Placebo
Drug: Varenicline — Participants will take one pill (.5 milligrams) a day for days 1-3 and then one pill (.5 milligrams) in the morning and one pill in the evening days 4-30 and months 2-12. In month 13 participants will take one pill in the morning days 1-3. Participants will be off study drug month 13 days 4-30.
  Other Names: Chantix
  Arms: Varenicline

SUMMARY:
This trial aims to test whether one year of Varenicline, when compared to placebo, can reduce fall risk and show improvement in the ability to multitask while walking.

Participants that are eligible after screening for the study will be randomized to receive Varenicline or placebo. Along with the study medication participants will have visits (over the phone and in person), various tests and imaging, questionnaires, and laboratory collections.

DETAILED DESCRIPTION:
The hypothesis of the trial are:

* The primary hypothesis is that varenicline will result in less progress in dual-task cost gait performance after 12 months of treatment compared to placebo in hypocholinergic Parkinson disease (PD) Mild Cognitive Impairment (MCI) patients.
* The primary secondary hypothesis assesses whether the magnitude of effect of varenicline relative to placebo is consistent with the minimal clinically important difference (MCID) for the relative risk of falls in the 12-month double-blind treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a PD diagnosis based on the Movement Disorders Society Clinical Diagnostic Criteria for Parkinson's Disease at the time of baseline screening/enrollment visit
* Participants with occipital association cortex cholinergic denervation in the lowest tertile of the normal range on F-fluoroethoxybenzovesamicol (FEOBV) Positron Emission Tomography (PET)
* Participants with legally authorized representatives (LARs) able to co-sign documented informed consent or participants that have capacity to provide informed consent upon study enrollment as ascertained by the study-specific University of California, San Diego Brief Assessment of Capacity to Consent (UBACC)
* Mild Cognitive Impairment consistent with Parkinson disease Mild Cognitive Impairment (PD-MCI)

Exclusion Criteria:

* Atypical Parkinsonian conditions other than Parkinson disease (PD)
* Participants initially on certain dopamine blocking drugs (per protocol), specific anticholinergic drugs (trihexyphenidyl, benztropine), or specific cholinesterase inhibitor drugs (per protocol) at the in-person screening visit
* Modified Hoehn and Yahr score of 4.0 or greater at the in-person screening visit
* Current or previous (within last 6 months of in-person screening visit) use of any product or medication containing nicotinic agents, including use of tobacco products such as cigarettes, cigars, pipes, chewing tobacco, etc., e-cigarettes, over the counter (OTC) nicotine patches, chewing gum containing nicotine, or varenicline
* Evidence of a stroke with both cortical and subcortical involvement or occipital lobe mass lesion on structural magnetic brain imaging (MRI) obtained at the in-person screening visit that would preclude co-registration and analysis of FEOBV PET data
* Participants where magnetic resonance imaging (MRI) is contraindicated including, but not limited to, those with a pacemaker, presence of metallic fragments near the eyes or spinal cord, or cochlear implant
* Severe claustrophobia precluding MRI or PET imaging
* Participants limited by participation in research procedures involving ionizing radiation
* Pregnancy (test within 48 hours of the PET imaging session in women of childbearing potential) or breastfeeding at the time of in-person screening visit
* Participants with stage 4 or 5 chronic kidney disease at the time of in-person screening visit (estimated Creatinine Clearance < 30 milliliters per minute)
* Current, significant mood disorder at the time of in-person screening/enrollment visit defined as follows: persistent (lasting longer than 2 weeks) symptoms of depression or anxiety in the 30 days preceding informed consent, as determined by self-report
* Evidence of active suicidal ideation as defined by an affirmative answer to either question 1 or 2 on the Columbia Suicide Severity Rating Scale (C-SSRS)
* History of a myocardial infarction or unstable angina in the 90 days preceding enrollment visit
* A current or previous history of epilepsy or any epileptic seizures in the 12 months preceding enrollment
* Heavy alcohol use as defined by a score of 8 or greater on the Alcohol Use Disorders Identification Test (AUDIT-self-report version) at the time of screening/enrollment visit
* Participants that are unable to swallow pills
* Participants with a history of allergic reaction to varenicline
* Participants that are actively taking part in another ongoing interventional (i.e., not observational) clinical trial

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2025-04-09 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Change in normal pace-dual task cost (npDTC) from baseline to 12 months. | Baseline, 12 months
  Normal pace-dual task cost is defined as the within-subject difference between normal pace walking speed without dual tasking to normal pace walking speed with dual tasking divided by normal pace walking speed without dual tasking, multiplied by 100.

SECONDARY OUTCOMES:
Number of falls from the first dose of study drug to the 12-month visit | First dose (day 0) to 12 month visit
  Participants will complete a fall diary to collect this data.

CONTACTS AND LOCATIONS:
Overall Officials: Vikas Kotagal, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
The study team will ensure the dataset is shared by the occurrence of the earlier of the following two milestones: either the date of primary publication or within 9 months of lifting of the data lock.
  De-identified subject data will be uploaded in a timely manner to a data repository using an established data transfer mechanism and the NINDS supported Common Data Elements (CDEs) as appropriate. Pending appropriate permissions, biospecimens (DNA) will be banked in the NINDS biorepository. Uploaded datasets will be coded and stripped of identifiers in order to prevent the possibility of identifying participants in this study from the publicly available dataset.
Supporting Information: Study Protocol, ICF
Time Frame: Access to the dataset that is uploaded to the data repository is available to any individual that applies to them for data access. This process does not place any limitations on the use of the data for commercial purposes.